CLINICAL TRIAL: NCT07092046
Title: How Safe is Minimal Flow Anesthesia in Terms of Infection?
Brief Title: Minimal Flow Anesthesia and Infection Risk
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Aysun ERŞEN YÜNGÜL, Specialist Physician, Ankara City Hospital Bilkent
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: EthicsApproval: E2-25-11471
Record Dates: First submitted 2025-07-20; First posted 2025-07-29 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Minimal Flow Anesthesia; General Anaesthesia; Inhalation Anesthesia; Infection Risk; Anesthesia Circuit; Microbial Colonization; Anesthesia Equipment Bacterial Contamination
Keywords: minimal flow anesthesia; Anesthesia Circuit; Infection Risk; Microbial Colonization
MeSH Terms: conditions — Communicable Diseases | interventions — Sevoflurane; Propofol; Remifentanil; Rocuronium; Sugammadex; Injections; Fentanyl; Atropine; Respiration, Artificial; Crystalloid Solutions; Intubation, Intratracheal

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Minimal Flow Anesthesia (0.5 L/min) (Active Comparator): Participants in this group will receive minimal-flow inhalation anesthesia, administered at a fresh gas flow rate of 0.5 L/min (Liters per minute). This technique helps preserve heat and humidity within the anesthesia circuit while reducing both anesthetic gas waste and environmental impact. The study aims to evaluate whether this lower flow rate contributes to circuit condensation and microbial colonization in the breathing system.
  Interventions: Drug: Sevoflurane (Volatile Anesthetic); Drug: Propofol 1%; Drug: Remifentanil 2 MG; Drug: Rocuronium 50 mg/5 ml; Drug: Lidocaine %2 ampoule; Drug: Ephedrine Hydrochloride 0,05 mg/ml ampoule; Drug: Sugammadex 200 MG in 2 ML Injection; Drug: Fentanyl (IV); Drug: Atropine Sulphate 0.5mg/ml ampoule; Procedure: Peripheral Intravenous Cannulation; Procedure: Mechanical Ventilation; Drug: Crystalloid solutions; Procedure: Endotracheal Intubation; Procedure: American Society of Anesthesiologists (ASA) Standard Monitors; Procedure: Minimal-Flow Anesthesia; Diagnostic Test: Anesthesia Circuit Sampling; Procedure: Body Temperature Monitoring; Diagnostic Test: Nasopharyngeal Swab Collection; Diagnostic Test: Microbiological Culture and Identification
- Standard Flow Anesthesia (2 L/min) (Active Comparator): Participants in this group will receive inhalation anesthesia with a continuous fresh gas flow rate of 2 liters per minute (L/min) throughout the surgical procedure. This represents conventional-flow anesthesia, in which higher gas turnover allows for rapid adjustments in anesthetic concentrations but may lead to increased loss of heat and humidity within the breathing circuit.
  Interventions: Drug: Sevoflurane (Volatile Anesthetic); Drug: Propofol 1%; Drug: Remifentanil 2 MG; Drug: Rocuronium 50 mg/5 ml; Drug: Lidocaine %2 ampoule; Drug: Ephedrine Hydrochloride 0,05 mg/ml ampoule; Drug: Sugammadex 200 MG in 2 ML Injection; Drug: Fentanyl (IV); Drug: Atropine Sulphate 0.5mg/ml ampoule; Procedure: Peripheral Intravenous Cannulation; Procedure: Mechanical Ventilation; Drug: Crystalloid solutions; Procedure: Endotracheal Intubation; Procedure: American Society of Anesthesiologists (ASA) Standard Monitors; Procedure: Normal-Flow Anesthesia; Diagnostic Test: Anesthesia Circuit Sampling; Procedure: Body Temperature Monitoring; Diagnostic Test: Nasopharyngeal Swab Collection; Diagnostic Test: Microbiological Culture and Identification

INTERVENTIONS:
Drug: Sevoflurane (Volatile Anesthetic) — An inhalational anesthetic agent will be used for the maintenance of anesthesia, administered at a concentration of 2-3% in a gas mixture consisting of 40% oxygen and air.
Drug: Propofol 1% — An intravenous hypnotic agent will be used for anesthesia induction at a dose of 2-3 mg/kg.
Drug: Remifentanil 2 MG — A short-acting opioid will be administered intravenously for maintenance of anesthesia at a dose of 0.02-0.2 micrograms per kilogram per minute (μg/kg/min).
Drug: Rocuronium 50 mg/5 ml — A neuromuscular blocking agent will be administered intravenously at a dose of 0.6-1.2 mg/kg for induction, and 0.15 mg/kg for maintenance of muscle relaxation during surgery.
Drug: Lidocaine %2 ampoule — This agent will be administered intravenously at a dose of 1-1.5 mg/kg prior to anesthesia induction to reduce injection pain and facilitate smooth induction.
Drug: Ephedrine Hydrochloride 0,05 mg/ml ampoule — This agent will be administered intravenously at a dose of 0.1 mg/kg to treat intraoperative hypotension that does not respond to fluid replacement or adjustment of anesthetic depth.
Drug: Sugammadex 200 MG in 2 ML Injection — Sugammadex will be administered intravenously at a dose of 2 mg/kg or 4 mg/kg, depending on the degree of neuromuscular blockade.
Drug: Fentanyl (IV) — Fentanyl will be administered intravenously as part of the anesthesia induction regimen, at a dose ranging from 1 to 2 micrograms per kilogram (µg/kg).
Drug: Atropine Sulphate 0.5mg/ml ampoule — In cases of intraoperative bradycardia, defined as a heart rate (HR) below 45 beats per minute (bpm), 0.5 mg of the agent will be administered intravenously.
Procedure: Peripheral Intravenous Cannulation — All participants received peripheral intravenous cannulation using 18-20 G IV cannulas placed on the dorsum of the hand before anesthesia induction.
Procedure: Mechanical Ventilation — Following endotracheal intubation, mechanical ventilation will be initiated using volume-controlled settings, with a tidal volume (TV) of 6-8 mL/kg, respiratory rate (RR) of 12 breaths per minute, and fraction of inspired oxygen (FiO₂) set at 50%. Ventilator parameters will be adjusted to maintain end-tidal carbon dioxide (ETCO₂) between 30 and 36 mmHg.
Procedure: Peripheral Intravenous Cannulation — All participants will undergo peripheral intravenous cannulation with 18-20 gauge (G) IV (intravenous) cannulas placed on the dorsum of the hand prior to anesthesia induction.
Drug: Crystalloid solutions — Participants will receive calculated maintenance fluid therapy with crystalloids administered via intravenous infusion, both prior to and throughout the surgical procedure.
Procedure: Endotracheal Intubation — Following induction of anesthesia and establishment of neuromuscular blockade, endotracheal intubation will be performed using a standard technique in all participants.
Procedure: American Society of Anesthesiologists (ASA) Standard Monitors — Routine monitoring in accordance with American Society of Anesthesiologists (ASA) guidelines, including noninvasive blood pressure, electrocardiogram (ECG, D2 lead), end-tidal carbon dioxide (ETCO₂), and peripheral oxygen saturation (SpO₂), will be performed in all patients starting from the preoperative period and continuing throughout the surgery.
Procedure: Minimal-Flow Anesthesia — In the minimal-flow anesthesia group, after induction and once a minimum alveolar concentration (MAC) of 1 is achieved, the fresh gas flow will be reduced to 0.5 L/min with a mixture of 45% oxygen (O₂) and 55% air, and maintained throughout the surgical procedure. At the end of surgery, the flow will be increased to 3 L/min to facilitate emergence. Disposable anesthesia circuits, bacterial filters, and face masks will be used for each patient, and carbon dioxide (CO₂) absorbers will be replaced daily.
  Arms: Minimal Flow Anesthesia (0.5 L/min)
Procedure: Normal-Flow Anesthesia — In the normal-flow anesthesia group, after induction and once a minimum alveolar concentration (MAC) of 1 is achieved, the fresh gas flow will be adjusted to 2 L/min and maintained during the surgical procedure. For emergence, the flow will be increased to 3 L/min. Disposable anesthesia circuits will be used, and daily maintenance protocols, including replacement of carbon dioxide (CO₂) absorbers, will be applied in the same manner as in the minimal-flow group.
  Arms: Standard Flow Anesthesia (2 L/min)
Diagnostic Test: Anesthesia Circuit Sampling — Sterile swab samples will be collected from both the inspiratory and expiratory limbs of the anesthesia circuit-once prior to circuit connection and again immediately after disconnection at the end of the surgical procedure. All samples will be processed for microbial culture and species-level identification.
Procedure: Body Temperature Monitoring — In addition to routine monitoring-including electrocardiogram (ECG), non-invasive blood pressure, peripheral oxygen saturation (SpO₂), and end-tidal carbon dioxide (ETCO₂)-body temperature will be continuously monitored in both study groups throughout the surgical procedure using appropriate thermal sensors. Temperature measurements will be recorded at 5-minute intervals and used to assess the impact of different fresh gas flow rates on intraoperative thermoregulation.
Diagnostic Test: Nasopharyngeal Swab Collection — A sterile nasopharyngeal swab (Dry SWAB) will be collected from each patient upon arrival in the operating room, prior to anesthesia induction. Each sample will be labeled with the patient's identification number, date, time, and collection site, and will be transferred in appropriate transport medium to the microbiology laboratory for culture and microbiological analysis.
Diagnostic Test: Microbiological Culture and Identification — All collected swab samples-including both nasopharyngeal and anesthesia circuit specimens-will be cultured using the serial dilution method on 5% sheep blood agar within 15 minutes of arrival at the microbiology laboratory. Cultures will be incubated at 35-37°C for 48 hours. Colony growth will be evaluated by a clinical microbiologist, and microorganisms will be identified to the species level using an automated MALDI-TOF MS (Matrix-Assisted Laser Desorption/Ionization Time-of-Flight Mass Spectrometry) system.

SUMMARY:
This study is being done to find out if the heat and moisture that build up during minimal flow anesthesia can lead to the growth of germs (microorganisms) inside the anesthesia equipment. Minimal flow anesthesia (using fresh gas flow of 0.5 liters per minute or less) is known to help protect the lungs and the environment. However, it may also cause water to collect in the equipment, which could allow germs to grow. In this study, we want to see whether this type of anesthesia is safe when it comes to the risk of germs in the equipment.

DETAILED DESCRIPTION:
Introduction Inhalation anesthesia is commonly administered using fresh gas flows between 2-6 L/min (liters per minute ). When this flow is reduced to 1 L/min, it is referred to as low-flow anesthesia, and when set at 0.5 L/min, it is known as minimal-flow anesthesia. The high-flow technique maintains a continuous supply of fresh gas within the system. However, since the patient inhales only a small portion of this gas, the majority is expelled into the anesthetic gas scavenging system. While this approach enables rapid adjustment of gas concentrations (O₂, anesthetic agents), the gases within the circuit remain cold and dry due to the removal of heat and humidity from the patient's lungs by soda lime. Additionally, a considerable amount of anesthetic gas is wasted.

In contrast, using fresh gas flows of ≤1 L/min decreases the amount of gas delivered from the vaporizers to the breathing circuit. This results in slower changes in gas concentrations but offers important advantages. Low-flow and minimal-flow anesthesia humidify and warm the inspired gases, which protect the patient's lungs. Compared to cold, dry gases, this improves mucociliary clearance, reduces damage to the respiratory epithelium, and lowers the release of inflammatory mediators. Low-flow anesthesia is a safe and effective practice that benefits patients and also provides economic and environmental advantages.

Minimal-flow anesthesia helps reduce heat loss through the respiratory tract and prevents the drying of mucosal surfaces, both of which are more common with higher flow rates. Additionally, it significantly decreases the amount of wasted fresh gas and inhaled anesthetic released into the atmosphere. Together, these effects may result in reduced airway inflammation and infection, lower environmental emissions, and cost savings.

Modern anesthesia machines support the safe delivery of low-flow anesthesia by utilizing closed breathing circuits that minimize leaks, manage humidity, ensure accurate gas delivery, and provide advanced monitoring and ventilator technologies.

Study Objective The primary objective of this study is to determine whether the increased humidity and temperature generated during minimal-flow anesthesia contribute to microbial colonization in the anesthesia circuit.

Methods A total of 140 patients undergoing elective surgical procedures will be included in this randomized, prospective, double-blind clinical trial. Eligible participants will be between 18 and 65 years of age, of either sex, and classified as ASA (American Society of Anesthesiologists) physical status I or II based on routine preoperative evaluation.

All participants will be informed about the study, including its objectives and potential risks, and written informed consent will be obtained. Patient demographics, including age, weight, ASA classification, and presence of chronic diseases, will be recorded prior to surgery. Randomization will be performed using the sealed envelope method.

Prior to each surgery, anesthesia circuits will undergo leak testing and gas monitor calibration. Disposable anesthesia circuits, bacterial filters, and masks will be used. The CO₂ absorbent (Sorbo-lime®, Berkim, Turkey) will be replaced daily. All anesthesia procedures will be performed using a GE Avance CS2 anesthesia machine. Standard intraoperative monitoring will include ECG (electrocardiogram ), non-invasive arterial blood pressure, SpO₂ (peripheral capillary oxygen saturation), respiratory rate, and ETCO₂ (End-tidal carbon dioxide). These parameters will be recorded at five-minute intervals. Body temperature monitoring will be added for study purposes.

Upon arrival in the operating room, nasopharyngeal swab samples will be collected under sterile conditions using dry sterile swabs (Dry SWAB) by trained personnel. All patients will undergo preoxygenation with 100% oxygen via face mask for three minutes at a fresh gas flow rate of 3 L/min during spontaneous ventilation. Anesthesia induction will be achieved using intravenous Lidocaine 1 mg/kg (milligrams per kilogram), Propofol 2 mg/kg, Fentanyl 1 mcg/kg (micrograms per kilogram), and Rocuronium 0.6-1 mg/kg, followed by endotracheal intubation.

Maintenance of anesthesia will be achieved using Sevoflurane to maintain MAC 1 (minimum alveolar concentration), along with a continuous Remifentanil infusion 0.02-0.2 mcg/kg/min (micrograms per kilogram per minute). Ventilator settings will include a tidal volume of 8 mL/kg (milliliters per kilogram), a respiratory rate of 12 breaths/min (minute), and an inspiratory-to-expiratory (I:E) ratio of 1:2. Anesthesia duration, vital parameters, body temperature, fresh gas flow settings, and ventilator settings will be recorded.

In both groups, fresh gas flow (O₂ 45%, Air 55%) will begin at 3 L/min. Once the MAC reaches 1, the flow rate will be reduced to 2 L/min in the normal-flow group and 0.5 L/min in the minimal-flow group. Ten minutes before the end of surgery, the fresh gas flow will be increased to 3 L/min in both groups, anesthetic agents will be discontinued, and 100% oxygen will be administered. Neuromuscular blockade will be reversed using Sugammadex 2-4 mg/kg, and patients will be extubated.

Swab samples will also be collected from the inspiratory and expiratory limbs of the disposable anesthesia circuits before connecting to the anesthesia machine and immediately after disconnection at the end of surgery-totaling four swabs per patient. All samples (nasopharyngeal and circuit swabs) will be labeled with the patient's name, date, site, and time of collection, then transported to the microbiology laboratory in a suitable transport medium at room temperature. Samples will be delivered to the laboratory within 15 minutes.

Microbiological analysis will be performed by inoculating the samples on 5% sheep blood agar using a dilution method. Incubation will be conducted at 35-37°C for 48 hours. Microbial growth will be assessed by a microbiologist, and species identification will be performed using an automated system (MALDI-TOF MS).

ELIGIBILITY:
Inclusion Criteria:

A total of 140 voluntary patients will be included in the study.

Patients will be aged between 18 and 65 years.

Both male and female patients will be enrolled.

All patients will be classified as c physical status I or II.

Patients will undergo elective surgical procedures.

The study will be conducted in the operating rooms of Ankara Bilkent City Hospital, affiliated with the Ministry of Health of the Republic of Türkiye.

-

Exclusion Criteria:

Patients who do not consent to participate

Patients outside the age range of 18-65 years

Patients classified as ASA (American Society of Anesthesiologists) III, IV, or V

Patients scheduled for emergency surgery

Patients with uncontrolled hypertension

Patients with significant cardiac diseases (e.g., heart failure, coronary artery disease, arrhythmia, valvular heart disease)

Patients with significant pulmonary diseases (e.g., Chronic Obstructive Pulmonary Disease, Restrictive Pulmonary Disease, Asthma)

Patients with neuromuscular disorders

Patients with poorly controlled diabetes mellitus

Patients with metabolic disorders

Patients with immunodeficiency

Patients with significant anemia

Patients with bleeding diathesis

Patients with liver and/or kidney diseases

History of cardiac surgery

History of intracranial surgery

History of pulmonary surgery

History of head and neck surgery

Anticipated difficult airway or difficult intubation

Patients with alcohol or drug dependence

Pregnant or lactating women

Known allergy to anesthetic agents

Body mass index (BMI) > 30 kg/m²

Presence of sepsis or active infection

Baseline body temperature < 35°C or > 38°C

Patients who have received antibiotics in the past month

Patients with malignancies

Withdrawal Criteria Patients who develop hemodynamic instability during the intraoperative period

Patients requiring interruption of minimal flow anesthesia for more than 5 minutes

Patients whose anesthesia circuit becomes disconnected intraoperatively

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of Bacterial Contamination in Anesthesia Circuits and Nasopharyngeal Swab Samples | During the observational period, which begins 10 minutes prior to anesthesia induction and continues until 10 minutes after the cessation of anesthesia.
  The aim of this study is to evaluate and compare bacterial contamination in the inspiratory and expiratory limbs of anesthesia circuits and in the nasopharyngeal region of patients undergoing elective surgery under either minimal-flow (0.5 L/min) or normal-flow (2 L/min) inhalation anesthesia. A total of four sterile swab samples will be collected from each patient: one nasopharyngeal swab upon arrival to the operating room, and three circuit swabs-two taken from the inspiratory and expiratory limbs before circuit connection, and one after circuit disconnection at the end of the procedure. All samples will be cultured and incubated under appropriate conditions, and microbial identification will be performed to the species level using matrix-assisted laser desorption/ionization time-of-flight mass spectrometry (MALDI-TOF MS).

SECONDARY OUTCOMES:
Changes in Body Temperature During Anesthesia | From 10 minutes before induction to 45 minutes after anesthesia termination
  Continuous body temperature monitoring will be conducted in all patients. Measurements will be recorded at 15-minute intervals, beginning 10 minutes prior to anesthesia induction and continuing until 45 minutes after the termination of anesthesia. The aim is to compare heart rate trends and perioperative variability between the two study groups: minimal-flow and normal-flow anesthesia.
Heart Rate at Defined Perioperative Time Points (bpm) | From 10 minutes before induction to 45 minutes after anesthesia termination
  Heart rate (HR) will be measured non-invasively using standard monitoring equipment in accordance with American Society of Anesthesiologists (ASA) guidelines. Measurements will be recorded at 15-minute intervals, beginning 10 minutes prior to anesthesia induction and continuing until 45 minutes after the termination of anesthesia. The objective is to compare heart rate trends and perioperative variability between the two study groups: minimal-flow and normal-flow anesthesia.
Peripheral Oxygen Saturation (SpO₂) at Defined Perioperative Time Points (%) | From 10 minutes before induction to 45 minutes after anesthesia termination
  Peripheral oxygen saturation (SpO₂) will be continuously monitored using pulse oximetry as part of standard monitoring in accordance with American Society of Anesthesiologists (ASA) guidelines. Measurements will be recorded at 15-minute intervals, beginning 10 minutes prior to anesthesia induction and continuing until 45 minutes after the termination of anesthesia. The objective is to compare heart rate trends and perioperative variability between the two study groups: minimal-flow and normal-flow anesthesia.
End-Tidal Carbon Dioxide (ETCO₂) Levels at Defined Perioperative Time Points (mmHg) | From 10 minutes before induction to 45 minutes after anesthesia termination
  End-tidal carbon dioxide (ETCO₂) will be continuously measured via the ventilator as part of standard intraoperative monitoring. Measurements will be recorded at 15-minute intervals, beginning 10 minutes prior to anesthesia induction and continuing until 45 minutes after the termination of anesthesia. The objective is to compare heart rate trends and perioperative variability between the two study groups: minimal-flow and normal-flow anesthesia.
Mean Arterial Pressure at Defined Perioperative Time Points (mmHg) | From 10 minutes before induction to 45 minutes after anesthesia termination
  Mean arterial pressure (MAP) will be measured non-invasively using standard monitoring equipment in accordance with American Society of Anesthesiologists (ASA) guidelines. Measurements will be recorded at 15-minute intervals, beginning 10 minutes prior to anesthesia induction and continuing until 45 minutes after the termination of anesthesia. The objective is to compare heart rate trends and perioperative variability between the two study groups: minimal-flow and normal-flow anesthesia.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Bilkent City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2023-03-20): https://cdn.clinicaltrials.gov/large-docs/46/NCT07092046/ICF_000.pdf